CLINICAL TRIAL: NCT04126252
Title: A Comparison of Pharmacotherapy and Psychotherapy in the Treatment of Erectile Dysfunction
Brief Title: Pharmacotherapy and Psychotherapy in the Treatment of Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Islamic University, Islamabad (Other)
Responsible Party: Principal Investigator, Ahmad Bilal, Principal Investigator, PhD Research Candidate, International Islamic University, Islamabad
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 0925-0586
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): This arm received pharmacotherapy for erectile dysfunction.
  Interventions: Drug: Sildenafil Citrate 50Mg Tab
- Group B (Experimental): This arm received cognitive behavior psychotherapy for erectile dysfunction.
  Interventions: Behavioral: Cognitive Behavioral Psychotherapy
- Group C (Experimental): This arm received combined treatment approach.
  Interventions: Combination Product: Combined or Integrated Therapy
- Group D (Placebo Comparator): This arm acted as a control group and received placebo or no intervention.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sildenafil Citrate 50Mg Tab — The Group A received sildenafil citrate 50 mg on demand for a period of max 3 months.
  Arms: Group A
Behavioral: Cognitive Behavioral Psychotherapy — The Group B received cognitive behavior psychotherapy for a period of max 3 months.
  Arms: Group B
Combination Product: Combined or Integrated Therapy — The Group C received the combined therapeutic approach for a period of max 3 months.
  Arms: Group C
Other: Placebo — The Group D received no treatment or placebo for a period of max 3 months.
  Arms: Group D

SUMMARY:
The study involved the administration of pharmacotherapy and cognitive behavior psychotherapy to individuals suffering from erectile dysfunction. The study was randomized controlled trial with four arms involving a control group.

ELIGIBILITY:
Inclusion Criteria:

* Men diagnosed with erectile dysfunction
* Must be in the age range of 18 to 40 years
* Must be in a stable heterosexual relationship
* Must not be suffering from any medical or psychiatric illness

Exclusion Criteria:

* Men not meeting criteria of diagnosis of erectile dysfunction
* Men not in a heterosexual relationship
* Men above the age of 40 years
* Men diagnosed with any medical or psychiatric illness

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Males
Enrollment: 116 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile Functioning-5 | 3 months maximum

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Bilal, Principal Investigator — International Islamic University, Islamabad, Pakistan
Locations (1):
- Ahmad Bilal Private Practice, Chak Four Hundred Fifty-four, Punjab Province, Pakistan

REFERENCES:
- [Derived] Bilal A, Abbasi NUH. Development of an indigenous manual of cognitive behavior sex therapy for young men. J Family Med Prim Care. 2022 Aug;11(8):4127-4130. doi: 10.4103/jfmpc.jfmpc_1892_21. Epub 2022 Aug 30. PMID 36353027